CLINICAL TRIAL: NCT01331265
Title: Understanding Perceived Lactose Intolerance in White, Black, and Hispanic Adults
Brief Title: Perceived Lactose Intolerance
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Theresa A Nicklas, Professor, Baylor College of Medicine
Other Study IDs: H-22651
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Lactose Intolerance
Keywords: perceived lactose intolerance; calcium/dairy consumption; specific health outcomes
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment

SUMMARY:
The goal of this study was to examine the effects of self-perceived lactose intolerance (SPLI) as it relates to calcium intake and specific health problems that have been attributed to reduced intake of calcium and foods from the dairy group in a nationally representative multi-ethnic sample of adults.

ELIGIBILITY:
Inclusion Criteria:

* adults between 18 and 50 years old

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: white, black, and Hispanic adults; 18-50 years of age
Sampling Method: Non-Probability Sample
Enrollment: 3815 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Nicklas TA, Qu H, Hughes SO, Wagner SE, Foushee R, Shewchuk RM. Prevalence of Self-reported Lactose Intolerance in a Multi-ethnic Sample of Adults. Nutrition Today 44(5):222-227, 2009
- [Result] Nicklas TA, Qu H, Hughes SO, He M, Wagner SE, Foushee HR, Shewchuk RM. Self-perceived lactose intolerance results in lower intakes of calcium and dairy foods and is associated with hypertension and diabetes in adults. Am J Clin Nutr. 2011 Jul;94(1):191-8. doi: 10.3945/ajcn.110.009860. Epub 2011 Apr 27. PMID 21525197